CLINICAL TRIAL: NCT05836038
Title: Creating Embodiment in Virtual Reality: A Pilot Study Evaluating Visio-tactile Stimulation and Feasibility
Brief Title: VR, Visio-tactile Stimulation and Embodiment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Nancy Baker, Associate Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM&E123
Record Dates: First submitted 2023-03-08; First posted 2023-05-01 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Virtual Reality; Visio-tactile stimulation; Feasibility; Embodiment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visio-tactile stimulation (VTS) during Virtual Reality (Experimental): Participants in this group will receive visio-tactile stimulation prior to engaging with the VR program. They will see their virtual hand touched while simultaneously feel their opposite real hand touched in the same pattern.
  Interventions: Behavioral: Visio-Tactile Stimulation
- No Visio-Tactile Stimulation (NoVTS) during Virtual Reality (No Intervention): Participants in this group will not receive visio-tactile stimulation prior to engaging with the VR program. They will be asked to look at their virtual hands for approximately the same amount of time as the VST group receive their stimulation

INTERVENTIONS:
Behavioral: Visio-Tactile Stimulation — They will see their virtual hand touched while simultaneously feel their opposite real hand touched in the same pattern.
  Arms: Visio-tactile stimulation (VTS) during Virtual Reality

SUMMARY:
Investigators will evaluate the feasibility of "puppeting" a virtual hand with the opposite hand in increasing complex movements and the effect of visio-tactile stimuli on embodiment to determine if it is a necessary part of the process.

DETAILED DESCRIPTION:
Embodiment refers to a subjective experience where a person views a simulated body and its properties are experienced as if they were the person's own biological body (1). Embodiment is notably seen in the rubber hand illusion (2): a rubber hand is made to substitute for the real hand using visio-tactile stimulation to connect the rubber hand to the participant. In visio-tactile stimulation, the real hand is hidden from view and the rubber hand is positioned where the real hand should be. Both hands are simultaneously stroked while the participant views the rubber hand. Within a short time, the rubber hand "feels" touch and pain, independent of the real hand.

In this study investigators will evaluate the ability to enable embodiment in a virtual reality environment. After providing background information, participants will then complete the "Real Hand Session" of the Study Protocol (See below) using their real hand to move the same side virtual hand (e.g. left real hand movements will move left virtual hand). Participants will complete Usability and Embodiment /Presence surveys After the Actual Protocol, participants in the VTS group will receive visio-tactile stimuli. They will see their virtual hand touched while simultaneously feel their opposite real hand touched in the same pattern. Participants in the NoVTS will spend the same amount of time looking at their virtual hand without the touching (~1 minute).

For the "Puppet Session" participants will complete the same tasks as the "Real Hand Session"(See Below) but movement of the real hand will "puppet" the opposite virtual hand (right real hand movements will move left virtual hand). After completing the session participants will complete Usability and Embodiment /Presence surveys

Study Protocol Sessions.(20 to 30 minutes). All take place in the virtual environment Hand Movement- Press a 36-button sequence 4x Bilateral Task - "Catch" 36 "fireflies" with both hands 4x. Unilateral Task - "Catch 36 "fireflies" with one hand 4x. Avoidance Task - Press a 36-button sequence. A "dangerous" virtual obstacle (e.g., sawblade) will be placed in the path of the virtual hand during some of the trajectories. Investigators will see how far from the most efficient trajectory participants moves to avoid the object

Hypotheses H1: Participants will demonstrate a greater sense of embodiment with visio-tactile stimuli (VTS) than without visio-tactile stimuli (NoVTS) H1a: Participants in the VTS group will report higher levels of embodiment than those in the NoVTS group.

H1b: Participants will demonstrate significantly better motor performance in the VTS group than the NoVTS group.

H1c: Participants in the VTS group will demonstrate greater avoidance of "dangerous items" than those in the NoVTS group H1d: Participants in the VTS group will report better usability of the embodied virtual hand than those in the NoVTS group.

H2: Motor Performance of the "Puppeted" virtual hand will be similar to the "Actual" virtual hand.

ELIGIBILITY:
Inclusion Criteria:

* • 30 adult participants (18+)

  * Right Handed

Exclusion Criteria:

* Seizure, loss of awareness, or other symptom linked to an epileptic condition in the last 5 years

  * Blind;
  * Unable to use hands to reach and grasp items
  * Implanted medical device such as a pacemaker, defibrillator, or hearing aid.
  * Contagious disorder on the face (such as pink eye) that could be transmitted via the VR head set or has open areas on the face or head that would come in contact with the headset;
  * Unable to understand and respond to English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Motor Performance - Speed | Through study completion, 1 day
  We will track and store participant movements during each task via the VR headset. These movements will be downloaded and processed to calculate speed
Motor Performance - Velocity | Through study completion, 1 day
  We will track and store participant movements during each task via the VR headset. These movements will be downloaded and processed to calculate velocity
Motor Performance - Precision | Through study completion, 1 day
  We will track and store participant movements during each task via the VR headset. These movements will be downloaded and processed to calculate Precision
Motor Performance - Trajectory | Through study completion, 1 day
  We will track and store participant movements during each task via the VR headset. These movements will be downloaded and processed to calculate trajectory
Motor Performance - Path Length | Through study completion, 1 day
  We will track and store participant movements during each task via the VR headset. These movements will be downloaded and processed to calculate path length
Motor Performance - Time to Target | Through study completion, 1 day
  We will track and store participant movements during each task via the VR headset. These movements will be downloaded and processed to calculate Time to target
Motor Performance - Error rate | Through study completion, 1 day
  We will track and store participant movements during each task via the VR headset. These movements will be downloaded and processed to calculate error rate
Embodiment | Through study completion, 1 day
  Participants perception of immersion during VR experience: Using Peck's Embodiment Scale (16 items scored on a 7 point likert scale with a final score between 1 and 7 with a higher score indicating greater emobidment) and the IPQ Presence questionnaire (14 items on a 7 point likert scale with a higher score indicating greater embodiment)
Presence | Through study completion, 1 day
  Participants perception of immersion during VR experience: IPQ Presence questionnaire (14 items on a 7 point likert scale with a score between 7 and 98 and a higher score indicating greater presence)
Usability - Engagement | Through study completion, 1 day
  Participants perception of the ease of use of the VR system using the User Engagement Scale (a 12 item 1-5 pt likert scale with scores between 12 and 60 and a higher score indicating greater usability)
Usability - Task Demands | Through study completion, 1 day
  Participants perception of the ease of use of the VR system using the NASA Task Index (6-item scored on 10 point VAS. Items are weighted by subject perception of what is important part of task. Higher score indicates greater task demand)
Usability - ease of use | Through study completion, 1 day
  Participants perception of the ease of use of the VR system using the System Usability Scale (10 item scored on 1-5 likert, scores are converted to a 100 scale with a higher score indicating greater ease of use)

IPD SHARING:
Plan to Share IPD: No